CLINICAL TRIAL: NCT05514626
Title: Three-dimensional (3D) Holographic Display for Ultrasound-Guided Structural Heart Disease Procedures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: RealView Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-14-001
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Structural Cardiac Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: 3D Holographic Display — 3D holographic visualization of the anatomy during the planned interventional procedure. The HOLOSCOPE-i will be used in addition to and will not replace conventional displays that are currently being used during the procedure.

SUMMARY:
This study is intended to evaluate the use of the holographic display of 3D images acquired during ultrasound based cardiac procedures and to assess the clinical use of the HOLOSCOPE-i, in providing 3D spatial understanding to the clinician performing the procedure. Patients scheduled to undergo an elective procedure in the Cardiac Catheterization Laboratory which use 3D echocardiography (ECHO) as part of the procedure will be enrolled to this study. In addition to the standard of practice imaging using ultrasound, patients anatomical structures will be evaluated using a 3D holographic system. The patients will complete their participation in the study, at the end of the procedure. No follow-up is required and patients will continue their routine medical care following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients are scheduled to undergo an elective procedure in the Cardiac Catheterization Laboratory which use 3D echocardiography (ECHO) as part of the procedure.

Exclusion Criteria:

* Denial of informed consent
* Any contraindications to three-dimensional echocardiographic imaging.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to Fifty (50) patients undergoing elective procedures which use 3D echocardiography for treatment of structural heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
HOLOSCOPE-i is of clinical use for ultrasound based cardiac procedures | During procedure
  Qualitative assessment using a Likert scale

SECONDARY OUTCOMES:
HOLOSCOPE-i provides an intuitive understanding of the spatial relationship of the anatomy | During procedure
  Qualitative assessment using a Likert scale
HOLOSCOPE-i provides an intuitive understanding of the spatial relationship between the tool and the anatomy | During procedure
  Qualitative assessment using a Likert scale
Satisfaction with the use of the HOLOSCOPE-i under intra-procedural conditions | During procedure
  Qualitative assessment using a Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No